CLINICAL TRIAL: NCT03569306
Title: Electromagnetic Navigation Bronchoscopy in the Diagnosis of Peripheral Pulmonary Nodules
Brief Title: ENB in the Diagnosis of Peripheral Pulmonary Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017YFC0112701-1
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Peripheral Pulmonary Nodules
Keywords: Electromagnetic navigation bronchoscopy(ENB); peripheral pulmonary nodules; diagnostic yield

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENB-EBUS-GS group (Experimental): ENB is used in this group.EBUS and GS are inserted into bronchi in the assistance of ENB. The EBUS probe and GS are confirmed to reach the lesion by EBUS images.
  Interventions: Device: ENB; Device: EBUS-GS
- EBUS-GS group (Active Comparator): ENB isn't used in this group.EBUS and GS are inserted into bronchi according to the chest CT that judged by the doctor. The EBUS probe and GS are confirmed to reach the lesion by EBUS images.
  Interventions: Device: EBUS-GS

INTERVENTIONS:
Device: ENB — ENB is carried out by a ENB system（LungCare, China) which can offer real-time navigation for bronchoscopy reaching peripheral pulmonary nodules.
  Arms: ENB-EBUS-GS group
Device: EBUS-GS — EBUS is performed using an endoscope ultrasound system , which is equipped with a 20-MHz mechanical radial-type probe (UM-S20-17S;Olympus) with an external diameter of 1.4 mm and a GS (K-201; Olympus).

SUMMARY:
The study is designed as a multi-center prospective trial with two arms, ENB-EBUS-GS group and EBUS-GS group, and aimed to evaluate the diagnostic yield and operation time between the two groups.

DETAILED DESCRIPTION:
The study is designed as a multi-center prospective trial with two arms, ENB-EBUS-GS group and EBUS-GS group, and aimed to evaluate the diagnostic yield and operation time between the two groups. Patients with peripheral pulmonary nodules that need to be confirmed by pathology will be enrolled in the study. A total of 400 patients are expected to be enrolled. EBUS will be used in both group. Biopsy, brushing and washing will be performed when EBUS image present. Brushing, washing and lavage will be performed when EBUS image absent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are older than 18 year-old.
2. Chest CT shows peripheral pulmonary nodule (8mm<longest diameter≤30mm) suspected to be malignant that need to be confirmed by pathology. The nodule is surrounded by lung parenchyma and invisible in standard bronchoscopy.
3. Patients who agree to undergo bronchoscopy without any contraindications.
4. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Chest CT scan shows that the pulmonary nodule is pure ground glass opacity.
2. Presence of concomitant endobronchial lesion during the brochoscopy procerdure.
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The difference of diagnostic yield between ENB-EBUS-GS group and EBUS-GS group | one year
  Diagnostic yield is defined as proportion of true positive and true negative.

SECONDARY OUTCOMES:
The difference of operation time between ENB-EBUS-GS group and EBUS-GS group | one week
  The operation time includes total operation time,total GS time and total EBUS time
The difference of complications between ENB-EBUS-GS group and EBUS-GS group | three months
  Complications mean a composite of operation-related serious adverse events (pneumothorax, bleeding, etc.) during and after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

REFERENCES:
- [Background] Gex G, Pralong JA, Combescure C, Seijo L, Rochat T, Soccal PM. Diagnostic yield and safety of electromagnetic navigation bronchoscopy for lung nodules: a systematic review and meta-analysis. Respiration. 2014;87(2):165-76. doi: 10.1159/000355710. Epub 2014 Jan 3. PMID 24401166
- [Background] Rivera MP, Mehta AC, Wahidi MM. Establishing the diagnosis of lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e142S-e165S. doi: 10.1378/chest.12-2353. PMID 23649436
- [Background] Seijo LM, de Torres JP, Lozano MD, Bastarrika G, Alcaide AB, Lacunza MM, Zulueta JJ. Diagnostic yield of electromagnetic navigation bronchoscopy is highly dependent on the presence of a Bronchus sign on CT imaging: results from a prospective study. Chest. 2010 Dec;138(6):1316-21. doi: 10.1378/chest.09-2708. Epub 2010 Apr 30. PMID 20435658
- [Background] Lamprecht B, Porsch P, Wegleitner B, Strasser G, Kaiser B, Studnicka M. Electromagnetic navigation bronchoscopy (ENB): Increasing diagnostic yield. Respir Med. 2012 May;106(5):710-5. doi: 10.1016/j.rmed.2012.02.002. Epub 2012 Mar 3. PMID 22391437
- [Background] Wang Memoli JS, Nietert PJ, Silvestri GA. Meta-analysis of guided bronchoscopy for the evaluation of the pulmonary nodule. Chest. 2012 Aug;142(2):385-393. doi: 10.1378/chest.11-1764. PMID 21980059
- [Derived] Zheng X, Cao L, Zhang Y, Xie F, Yang H, Liu J, Qu S, Zhang J, Sun J. A Novel Electromagnetic Navigation Bronchoscopy System for the Diagnosis of Peripheral Pulmonary Nodules: A Randomized Clinical Trial. Ann Am Thorac Soc. 2022 Oct;19(10):1730-1739. doi: 10.1513/AnnalsATS.202109-1071OC. PMID 35679184